CLINICAL TRIAL: NCT06038539
Title: A Multicenter, Double-blind, Randomized, Parallel-group, Phase 3 Study to Compare the Efficacy and Safety of the Proposed Biosimilar PERT-IJS and EU-Perjeta® Along With Trastuzumab and Chemotherapy (Carboplatin and Docetaxel) as Neoadjuvant Treatment in Patients With Hormone Receptor Negative (HR-ve) Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Early Stage or Locally Advanced Breast Cancer
Brief Title: Efficacy and Safety of the Proposed Biosimilar Pertuzumab (PERT-IJS) Versus EU-Perjeta® Along With Trastuzumab and Chemotherapy (Carboplatin and Docetaxel) as Neoadjuvant Treatment in Chemotherapy naïve Patients With Early Stage or Locally Advanced HR Negative and HER2 Positive Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocon Biologics UK Ltd (Industry)
Responsible Party: Sponsor
Organization: Biocon Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-PERTUZ-301
Record Dates: First submitted 2023-08-23; First posted 2023-09-15 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: HR Negative HER2 Positive Early Breast Cancer or Locally Advanced Breast Cancer Patients
Keywords: Locally advanced breast cancer patient; HR negative HER2-positive Early breast cancer; PERT-IJS; Pertuzumab; Trastuzumab; Neoadjuvant treatment
MeSH Terms: interventions — Trastuzumab; Carboplatin; Docetaxel; pertuzumab

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A: PERT-IJS plus trastuzumab, carboplatin and docetaxel (Experimental): Part 1 (Cycle 1 to 6):
  Initial loading dose of PERT-IJS is 840 mg administered as an approximately 60-minute IV infusion followed every 3 weeks by a maintenance dose of 420 mg administered as an IV infusion over a period of approximately 30 to 60 minutes.
  Trastuzumab: Initial dose of trastuzumab is 8 mg/kg administered as approximately 90-minute IV infusion followed every 3 weeks by 6 mg/kg IV infusion over 30 to 90 minutes Carboplatin: Area Under the Curve (AUC) 6 for Cycles 1 to 6 Docetaxel: 75 mg/m2 by IV infusion every 3 weeks for Cycles 1 to 6
  Part 2 (Cycle 7 - till end of 1 year from Cycle 1 day 1):
  Initial loading dose of PERT-IJS is 840 mg administered as approximately 60-minute IV infusion followed every 3 weeks by a maintenance dose of 420 mg administered as an IV infusion over a period of approximately 30 to 60 minutes.
  Trastuzumab: As mentioned in part 1
  Interventions: Biological: PERT-IJS plus trastuzumab, carboplatin and docetaxel
- Treatment Arm B: EU-Perjeta plus trastuzumab, carboplatin and docetaxel (Active Comparator): Part 1 (Cycle 1 to 6):
  Initial loading dose of EU- Perjeta is 840 mg administered as approximately 60-minute IV infusion followed every 3 weeks by a maintenance dose of 420 mg administered as an IV infusion over a period of approximately 30 to 60 minutes.
  Trastuzumab: Initial dose of trastuzumab is 8 mg/kg administered as approximately 90-minute IV infusion followed every 3 weeks by 6 mg/kg IV infusion over 30 to 90 minutes Carboplatin: Area under the curve 6 for Cycles 1 to 6 Docetaxel: 75 mg/m2 by IV infusion every 3 weeks for Cycles 1 to 6
  Part 2 (Cycle 7 onwards till end of 01 year from Cycle 1 day 1):
  The patients will be re-randomized (1:1) to receive EU- Perjeta + trastuzumab or PERT-IJS + trastuzumab.
  Initial loading dose of PERT-IJS is 840 mg administered as approximately 60-minute IV infusion followed every 3 weeks by a maintenance dose of 420 mg administered as an IV infusion over a period of approximately 30 to 60 minutes.
  Trastuzumab: As mentioned in part 1
  Interventions: Biological: Perjeta plus trastuzumab, carboplatin and docetaxel

INTERVENTIONS:
Biological: PERT-IJS plus trastuzumab, carboplatin and docetaxel — PERT-IJS is a monoclonal antibody, which has been developed by Biocon Biologics (earlier in collaboration with Viatris) as a proposed biosimilar to European Union (EU)-approved and United States (US) licensed Perjeta.
  Arms: Treatment Arm A: PERT-IJS plus trastuzumab, carboplatin and docetaxel
Biological: Perjeta plus trastuzumab, carboplatin and docetaxel — EU Perjeta (Pertuzumab) , an antineoplastic agent, is a recombinant humanized monoclonal antibody that specifically targets sub-domain 2 of the extracellular domain of Human Epidermal Growth Factor Receptor 2 (HER2), blocking heterodimerization of HER2 with other members of the receptor family, including epidermal growth factor, Human Epidermal Growth Factor Receptor 3 (HER3) and Human Epidermal Growth Factor Receptor 4 (HER4).
  Arms: Treatment Arm B: EU-Perjeta plus trastuzumab, carboplatin and docetaxel

SUMMARY:
To compare the efficacy and safety of PERT-IJS (Proposed biosimilar Pertuzumab) plus trastuzumab and chemotherapy (carboplatin and docetaxel) versus EU-Perjeta plus trastuzumab and chemotherapy (carboplatin and docetaxel) in neoadjuvant treatment of patients with HR-ve and HER-2 positive early stage or locally advanced breast cancer.

DETAILED DESCRIPTION:
This study is designed to compare the efficacy and safety of proposed biosimilar PERT-IJS plus trastuzumab, carboplatin and docetaxel versus EU-Perjeta plus trastuzumab, carboplatin and docetaxel in neoadjuvant treatment of HR-ve HER2-positive Early Breast Cancer (EBC) (invasive breast cancer without distant metastasis) or locally advanced breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient willing and able to sign informed consent and to follow the protocol requirements
2. Female patients aged ≥ 18 years at the time of Screening
3. Patient with Eastern Cooperative Oncology Group (ECOG) Performance Status < 2
4. Patients with breast cancer that meets the following criteria:

   1. A known case of histologically confirmed invasive breast carcinoma with a primary tumor size of > 2 cm by standard local assessment technique
   2. stage at presentation: early stage (T2-3, N0-1, M0) or locally advanced (T2-3, N2 or N3, M0; T4a-c, any N, M0) or inflammatory (T4d, any N, M0)
5. Patients with HER2 overexpression by Immunohistochemistry (IHC) (defined as IHC 3+, or IHC 2+ with Fluorescence In Situ Hybridization (FISH) confirmation) as per the American Society of Clinical Oncology/College of American Pathologist (ASCO-CAP) guidelines prior to Screening and confirmed centrally before randomization
6. Patients with known HR-ve status (ER-negative and PR-negative) as per local laboratory prior to Screening and confirmed centrally before randomization
7. Patient willing to undergo mastectomy or breast-conserving surgery after neoadjuvant therapy
8. Patient who completes all necessary baseline laboratory and radiologic investigations prior to randomization as per Schedule of assessment (SoA)
9. Patient with baseline left ventricular ejection fraction (LVEF) ≥ 55% measured by echocardiography (ECHO; preferred) or multiple-gated acquisition (MUGA) scan
10. Patient is eligible to participant if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

Exclusion Criteria:

1. Patients with metastatic or recurrent bilateral breast cancer, or bilateral breast cancer
2. Patients with a history of concurrent or previously treated non-breast malignancies. A patient with previous invasive non-breast cancer is eligible provided she has been disease free for more than 5 years
3. Patients who have received any previous systemic therapy (including chemotherapy, immunotherapy, HER2-targeted agents, and antitumor vaccines) for treatment or prevention of breast cancer, or radiation therapy for treatment of cancer
4. Concurrent anti-cancer treatment in another investigational study, including hormone therapy or immunotherapy
5. Major surgical procedure that is unrelated to breast cancer within 4 weeks prior to randomization or from which the patient has not fully recovered
6. Serious cardiac illness or medical condition including but not limited to the following as per Investigator's discretion:

   1. Patients with ≥ Class II stage of heart failure as per New York Heart Association Classification
   2. High risk uncontrolled arrhythmia, such as atrial tachycardia with a heart rate > 100 bpm at rest, significant ventricular arrhythmia (e.g., ventricular tachycardia) required treatment, or higher-grade atrioventricular (AV) block (i.e., Mobitz II second-degree AV block or third-degree AV block)
   3. History of myocardial infarction or unstable angina pectoris within 1 year of randomization or angina pectoris requiring anti-anginal medication
   4. Evidence of transmural infarction on ECG
   5. Clinically significant valvular heart disease
   6. Poorly controlled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg) in patients on anti-hypertensive medications
7. Other concurrent serious diseases that may interfere with study primary endpoint and other study assessments, including, but not limited to, severe pulmonary conditions/illness, active liver disease (for example, active viral hepatitis infection [i.e., hepatitis B or hepatitis C]), autoimmune disorders, history of or known patient of sclerosing cholangitis, or infection with Human immune deficiency virus (HIV)
8. Patients with a history of any contraindication to the study treatment regimens
9. Any of the following abnormal laboratory test results prior to randomization:

   1. Total bilirubin > upper limit of normal (ULN) or, for cases of known Gilbert's syndrome, total bilirubin > 2 × ULN
   2. Aspartate aminotransferase and/or alanine aminotransferase > 1.5 × ULN, if considered clinically significant by Investigator
   3. Alkaline phosphatase >2.5 × ULN, if considered clinically significant by Investigator
   4. Serum creatinine > 1.5 × ULN
   5. Creatinine clearance < 60 mL/min
   6. Total white blood cells count < 2500 cells/μL
   7. Absolute neutrophil count < 2000 cells/μL
   8. Platelet count < 100,000 cells/μL
10. Participation in any clinical study with an investigational drug, biologic, or device within 1 month prior or within five half-lives (of the drug/ biologic) prior to the enrolment (whichever is longer)
11. Have taken any live vaccines 30 days prior to the 1st dose of study treatment
12. Any known hypersensitivity to any of the study medications, any of the ingredients or excipients of these medications, or benzyl alcohol
13. Patients unwilling to follow the study requirements.
14. Presence of an uncontrolled, unstable, clinically significant medical condition that, in the opinion of the Investigator, may interfere with the interpretation of efficacy and safety parameters or has a medical condition for which the treatment should take precedence over study participation or will interfere with study participation

    -

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 382 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint - Total pathologic complete response between Treatment arm A and Treatment Arm B | Week 18
  Total pathologic complete response (tpCR; ypT0/Tis,ypN0) in breast and axillary nodes after neoadjuvant treatment by Independent Review Committee (IRC)

SECONDARY OUTCOMES:
Efficacy endpoint-Total pathologic complete response between Treatment Arm A and Treatment Arm B as neoadjuvant treatment regimen | Week 18
  Total pathologic complete response (tpCR; ypT0/Tis, ypN0) in breast and axillary nodes after neoadjuvant treatment by local histopathologist
Efficacy endpoint: Pathologic complete response between Treatment Arm A and Treatment Arm B | Week 18
  Pathologic complete response (pCR; ypT0/ypN0) after neoadjuvant treatment by IRC and local histopathologist
Efficacy endpoint- Breast pathologic complete response between Treatment Arm A and Treatment Arm B as neoadjuvant treatment regimen | Week 18
  Breast pathologic complete response (bpCR; ypT0/Tis) after neoadjuvant treatment by IRC and local histopathologist
Efficacy endpoint-Objective response rate between Treatment Arm A and Treatment Arm B as neoadjuvant treatment regimen | Week 18
  Objective response rate (ORR) after neoadjuvant treatment in accordance with Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
Efficacy endpoint-Event free survival rate between Treatment Arm A and Treatment Arm B as neoadjuvant treatment regimen | Week 18
  Event free survival (EFS) rate
Efficacy endpoint- Overall survival rate between Treatment Arm A and Treatment Arm B as neoadjuvant treatment regimen | Week 18
  Overall survival (OS) rate
Efficacy endpoint-EFS rate of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta throughout | 1 Year
  EFS rate
Efficacy endpoint - Overall Survival rate of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta throughout | 1 Year
  Overall survival rate
Efficacy endpoint - Overall Response Rate of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta throughout | 1 Year
  Overall Response Rate
Efficacy Endpoint: EFS rate after the single switch from EU-Perjeta to PERT-IJS+trastuzumab compared with those continuing on Treatment B | 1 year
  EFS rate after switching of treatment from EU-Perjeta to PERT-IJS + trastuzumab
Efficacy Endpoint: Disease free survival rate after the single switch from from EU-Perjeta to PERT-IJS+trastuzumab compared with those continuing on EU-Perjeta+trastuzumab | 1 year
  Disease free survival (DFS) rate after switching of treatment from EU-Perjeta to PERT-IJS + trastuzumab versus those continuing on EU-Perjeta + trastuzumab
Efficacy Endpoint: Overall survival rate after the single switch from from EU-Perjeta to PERT-IJS+trastuzumab compared with those continuing on EU-Perjeta+trastuzumab | 1 year
  OS rate after switching of treatment from EU-Perjeta to PERT-IJS + trastuzumab versus those continuing on EU-Perjeta + trastuzumab
Pharmacokinetic (PK) endpoint-The trough serum concentration | 1 Year
  The trough serum concentration (Ctrough)
Safety Endpoint: treatment-emergent adverse events and serious adverse events | week 18
  Incidence and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)
Safety Endpoint: left ventricular ejection fraction | week 18
  Incidence of patients with a decline in left ventricular ejection fraction (LVEF) of ≥ 10% from baseline to < 50%
Safety Endpoint: Vital signs | week 18
  Number of subjects with clinically significant changes in Vital signs
Safety Endpoint-ECG PR Interval | week 18
  Number of subjects with clinically significant changes in ECG PR Interval
Safety Endpoint-ECG QRS Interval | week 18
  Number of subjects with clinically significant changes in ECG QRS Interval
Safety Endpoint-ECG QT Interval | week 18
  Number of subjects with clinically significant changes in ECG QT Interval
Safety Endpoint- ECG corrected QT interval (QTc) Interval | week 18
  Number of subjects with clinically significant changes in ECG QTc Interval
Safety Endpoint-clinical laboratory assessments | week 18
  Number of subjects with clinically significant changes in Clinical laboratory assessments
Safety Endpoint-pregnancy test | week 18
  Number of subjects with Pregnancy outcome
Safety Endpoint-physical examination | week 18
  Number of subjects with clinically significant changes in Physical examination
Immunogenicity Endpoint | week 18
  Immunogenicity (anti-drug antibodies (ADA) and neutralizing antibodies (nAb) titers)
Safety Endpoint: treatment-emergent adverse events and serious adverse events of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta | 1 year
  Incidence and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)
Safety Endpoint: left ventricular ejection fraction of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta throughout | 1 year
  Incidence of patients with a decline in left ventricular ejection fraction (LVEF) of ≥ 10% from baseline to < 50%
Safety Endpoint: Routine safety parameters of patients randomized to PERT-IJS -throughout compared to patients randomized to EU-Perjeta throughout- Vital signs | 1 year
  Number of subjects with clinically significant changes in Vital signs
Safety Endpoint: Routine safety parameters of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta throughout- ECG PR Interval | 1 year
  Number of subjects with clinically significant changes in ECG PR Interval
Safety Endpoint: Routine safety parameters of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta throughout-ECG QRS Interval | 1 year
  Number of subjects with clinically significant changes in ECG QRS Interval
Safety Endpoint: Routine safety parameters of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta throughout-ECG QT Interval | 1 year
  Number of subjects with clinically significant changes in ECG QT Interval
Safety Endpoint: Routine safety parameters of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta throughout- ECG QTc Interval | 1 year
  Number of subjects with clinically significant changes in ECG QTc Interval
Safety Endpoint: Routine safety parameters of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta throughout-Clinical laboratory assessments | 1 year
  Number of subjects with clinically significant changes in Clinical laboratory assessments
Safety Endpoint: Routine safety parameters of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta throughout- Pregnancy test | 1 year
  Number of subjects with Pregnancy outcome
Safety Endpoint: Routine safety parameters of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta throughout-Physical examination | 1 year
  Number of subjects with clinically significant changes in Physical examination
Immunogenicity Endpoint of patients randomized to PERT-IJS throughout compared to patients randomized to EU-Perjeta throughout | 1 year
  Immunogenicity (anti-drug antibodies (ADA) and neutralizing antibodies (nAb) titers)
Safety Endpoint: Incidence of TEAEs and SAEs after the single switch from EU-Perjeta to PERT-IJS+trastuzumab versus those continuing on EU-Perjeta+trastuzumab throughout | 1 Year
  Incidence of TEAEs and SAEs after switching of treatment from EU-Perjeta to PERT-IJS + trastuzumab versus those continuing on EU-Perjeta + trastuzumab
Safety End Point :left ventricular ejection fraction incidences after the single switch from EU-Perjeta to PERT-IJS+trastuzumab versus those continuing on EU-Perjeta+trastuzumab | 1 year
  Incidence of patients with a decline in left ventricular ejection fraction (LVEF) of ≥ 10% from baseline to < 50%
Immunogenicity End Point: after the single switch from EU-Perjeta to PERT-IJS+trastuzumab versus those continuing on EU-Perjeta+trastuzumab | 1 Year
  Immunogenicity (ADA titer and nAb titer) after switching of treatment from EU-Perjeta to PERT-IJS plus trastuzumab versus those continuing on EU-Perjeta + trastuzumab

CONTACTS AND LOCATIONS:
Locations (1):
- Chopda Medicare & Research Centre Pvt. Ltd,, Nashik, India

IPD SHARING:
Plan to Share IPD: No